CLINICAL TRIAL: NCT02565758
Title: A Multicenter, Phase 1, Open-Label, Dose-Escalation Study of ABBV-085, an Antibody Drug Conjugate, in Subjects With Advanced Solid Tumors
Brief Title: ABBV-085, an Antibody Drug Conjugate, in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-394; 2015-001645-84 (EudraCT Number)
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Advanced Solid Tumors; Undifferentiated Pleomorphic Sarcoma; Squamous Cell Carcinoma of the Head and Neck; Carcinoma of the Breast
Keywords: Cancer; Advanced Solid Tumors; Neoplasm; Undifferentiated pleomorphic sarcoma; squamous cell carcinoma of the head and neck; carcinoma of the breast; antibody drug conjugate
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A4 (ABBV-085) (Experimental): ABBV-085 administered on at 28 day cycle and enrolling at MD Anderson
  Interventions: Drug: ABBV-085
- Arm A3 (ABBV-085) (Experimental): ABBV-085 will be administered at every cycle (28-day cycles).
  Interventions: Drug: ABBV-085

INTERVENTIONS:
Drug: ABBV-085 — Administered as an intravenous infusion in 28-day dosing cycles.

SUMMARY:
This is an open-label dose escalation study designed to evaluate the safety and pharmacokinetics of ABBV-085 and determine the recommended Phase 2 dose (as monotherapy or in combination with standard therapies) in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with advanced solid tumor that is not amenable to surgical resection or other approved therapeutic options.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
3. Participants must have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or disease evaluable by assessment of tumor antigens:

   - Participants with non-evaluable or non-measurable cancer are eligible if they have a confirmed increase in tumor antigens >=2 x upper limit of normal (ULN).
4. All participants must consent to provide archived diagnostic formalin-fixed paraffin embedded (FFPE) tumor tissue and on study biopsies.
5. Participant has adequate bone marrow, renal, hepatic and cardiac function.
6. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment.

Exclusion Criteria:

1. Participant has received anticancer therapy or any investigational therapy within a period of 21 days prior to the first dose of ABBV-085.
2. Uncontrolled metastases to the central nervous system (CNS). Participants with brain metastases are eligible provided they have shown clinical and radiographic stable disease for at least 4 weeks after definitive therapy and have not used steroids for at least 4 weeks prior to first dose of ABBV-085.
3. Unresolved adverse events >= Grade 2 from prior anticancer therapy, except for alopecia.
4. Participant has ongoing hemolysis.
5. Major surgery within <=28 days prior to the first dose of ABBV-085.
6. Clinically significant uncontrolled condition(s).
7. Participant has history of major immunologic reaction to any auristatin-based and /or Immunoglobulin G (IgG) containing agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Terminal elimination half life of ABBV-085. | UP to 24 months
Maximum observed plasma concentration (Cmax) of ABBV-085. | Up to 24 months
Number of participants with Adverse Events | Up to 24 months
  Collect all adverse events at each visit.
Area under the curve (AUC) from time zero to the last measurable concentration AUC(0-t) of ABBV-085. | Up 24 months
  AUC (0-t) = Area under the serum concentration curve from time zero (pre-dose) to the time of the last measurable concentration.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months
  ORR is defined as the proportion of the participants who achieve a complete response (CR) or partial response (PR).
Progression free survival (PFS) | Up to 24 months
  PFS is defined as the time from the first dose date of ABBV-085 to either disease progression or death, whichever occurs first.
Duration of overall response (DOR) | Up to 24 months
  DOR is defined as the time from the participant's initial CR or PR to the time of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (20):
- United States (16):
  - Mayo Clinic Arizona /ID# 148582, Phoenix, Arizona
  - Scottsdale Healthcare /ID# 151349, Scottsdale, Arizona
  - University of California, Los Angeles /ID# 148586, Los Angeles, California
  - Univ of Colorado Cancer Center /ID# 148581, Aurora, Colorado
  - University of Chicago /ID# 148579, Chicago, Illinois
  - Dana-Farber Cancer Institute /ID# 143782, Boston, Massachusetts
  - Washington University-School of Medicine /ID# 151348, St Louis, Missouri
  - NYU Langone Medical Center /ID# 150786, New York, New York
  - Duke Univ Med Ctr /ID# 148200, Durham, North Carolina
  - Carolina BioOncology Institute /ID# 148583, Huntersville, North Carolina
  - University of Pennsylvania /ID# 148576, Philadelphia, Pennsylvania
  - Greenville Hospital System /ID# 148652, Greenville, South Carolina
  - Mary Crowley Cancer Research /ID# 148580, Dallas, Texas
  - Univ TX, MD Anderson /ID# 147681, Houston, Texas
  - South Texas Accelerated Research Therapeutics /ID# 141715, San Antonio, Texas
  - Virginia Cancer Specialists /ID# 148584, Fairfax, Virginia
- Gustave Roussy /ID# 150300, Villejuif, Île-de-France Region, France
- Spain (3):
  - Hospital Univ Ramon y Cajal /ID# 150799, Madrid
  - Fundacion Jimenez Diaz /ID# 148564, Madrid
  - Hosp Univ Madrid Sanchinarro /ID# 146039, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ray U, Pathoulas CL, Thirusangu P, Purcell JW, Kannan N, Shridhar V. Exploiting LRRC15 as a Novel Therapeutic Target in Cancer. Cancer Res. 2022 May 3;82(9):1675-1681. doi: 10.1158/0008-5472.CAN-21-3734. PMID 35260879